CLINICAL TRIAL: NCT02387047
Title: Screening for Phobia of Falling in the Elderly: Validity and Feasibility of a Self-administered Questionnaire
Brief Title: Validity of a Self-administered Questionnaire to Screen Phobia of Falling in the Elderly
Acronym: PACTE-q
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 14SDE-PACTEQ
Record Dates: First submitted 2015-01-27; First posted 2015-03-12 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Phobic Disorders
MeSH Terms: conditions — Phobic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to determine the validity of a self-questionnaire detecting seniors phobia of falling living at home. A prospective monocentric observational study compares in a blind way the presence of Diagnostic and Statistical Manual of Mental Disorders fourth edition (DSM-IV) criteria for specific phobia, considered as the gold standard to the score obtained at the detecting questionnaire for ≥70 years old seniors suspected of phobia of falling and attending geriatric day hospital at the Bretonneau hospital (APHP, Paris).

DETAILED DESCRIPTION:
Context : The phobia of falling strongly contributes to the frailty of the elderly, and plays a key role in falls occuring and their deleterious effect. It concerns a big part of seniors living at home, fell before or not, and frequently leads to a restriction of their mobility. When the phobia of falling occurs, the fear of falling down takes an excessive scope, it is associated with anxious reactions when seniors dread the risk, and leads them to avoid these situations reducing their mobility. This reduction of activities contributes to the premature decline of physical capacities, worsens social life, increases the falling and institutionalization risk. However, there is no specific tools for the detection of seniors falling phobia, enabling us to turn patients towards a therapeutic and diagnostical adapted care. A detecting self-questionnaire was thus designed by the research geriatric team after an analysis of the literature and half-directive interviews with a representative sample of the target population.

Objectives : The main objective of this study is to evaluate the validity of a self-questionnaire so as to detect falling phobic seniors living at home. The optimal threshold of the questionnaire score, obtained from a receiver operating characteristic curve (ROC curve), will let us evaluate its concordance compared to the gold standard, formed by DSM-IV criteria for specific phobia. The results of the questionnaire will be kept secret while the study occurs. The secondary objectives will be to control the feasibility of the self-questionnaire detecting phobia of falling, the validity of internal structure and external construction by the exploration of its correlation with other close psychological and physical health measures.

Design : A 1 year prospective monocentric observational study is led with seniors attending geriatric day hospital at the Bretonneau hospital (APHP, Paris). While the same day hospital, all eligible patients will have a current evaluation of cares adapted to their admission causes. These patients will fill out the self-questionnaire detecting phobia, designed by the research geriatric team. The final clinical diagnostic of phobia of falling will be disconfirmed or affirmed from DSM-IV-TR (TR stands for text revision) criteria. At the end of the day hospital, an adapted care to their pathologies will be suggested to all the patients, according to usual practice.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years and over
* Presenting walking difficulties and/or disturbance of the balance and/or at least one fall during the course of the last 5 years and/or a fear of falling
* Living in community
* Non opposition of the patient to the collection of his personal data

Exclusion Criteria:

* Depression
* Cognitive disorders
* Inability to communicate

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Consecutive patients aged 70 years or more, consulting in geriatric day hospital, presenting walking difficulties and/or disturbance of the balance and/or at least one fall during the course of the last 5 years and/or a fear of falling, living in community
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Concordance of the self-questionnaire score compared to the gold standard formed by DSM-IV criteria for specific phobia presence | 1 day
  In a first time, the optimal threshold of the self-questionnaire score will be determined with a ROC curve. In a second time, this threshold will let us evaluate the score concordance compared to reference method.

SECONDARY OUTCOMES:
Percentage of filled out self-questionnaires | 1 day
  Evaluation of construct validity of the self-questionnaire
Item response rate | 1 day
  Evaluation of construct validity of the self-questionnaire
Help requirement to fill out the self-questionnaire | 1 day
  Evaluation of construct validity of the self-questionnaire
Time to complete the self-questionnaire | 1 day
  Evaluation of construct validity of the self-questionnaire
Patients' satisfaction with the self-questionnaire | 1 day
  Evaluation of construct validity of the self-questionnaire
Life-space mobility assessed by the Life-Space Assessment | 1 day
Comorbidity assessed by the Cumulative Illness Rating Scale for Geriatrics | 1 day
History of falls, number and gravity | 1 day
Frailty assessment according to phenotype definition of Fried | 1 day
  Evaluation of construct validity of the self-questionnaire
The Fear Questionnaire | 1 day
The Mobility Inventory for Agoraphobia | 1 day
Fear of falling assessed by the Falls Efficacy Scale-International | 1 day
Self-rated health assessed by the Minimum European Health Module | 1 day
The Timed Up and Go, performance-Oriented Mobility Assessment, 10-m walk test, the 30-s chair-stand test | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Delpierre, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bretonneau, Paris, France